CLINICAL TRIAL: NCT06736795
Title: Progressive Achilles Loading Via Clinician E-support (PACE)
Brief Title: Progressive Achilles Loading Via Clinician E-support
Acronym: PACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruth Chimenti (Other)
Collaborators: C.R.Darnall Army Medical Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ruth Chimenti, Associate Professor, Physical Therapy and Rehabilitation Science, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202405285; HT94252410536 (Other Grant/Funding Number: US Department of Defense, Congressionally Directed Medical Research Programs (CDMRP-PRORP))
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Achilles Tendon Pain; Achilles Tendinopathy
Keywords: ultrasound imaging; tendon health; pain; exercise; physical therapy; education
MeSH Terms: conditions — Pain; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-visit, Physical Therapist Initiated and Self-Pace Rehabilitation (Experimental): Participants will complete 6 online modules, which will take 10 to 20 minutes each. The modules can be completed at their own pace over 8 weeks and include:
  1. Exercise participation: Participants will receive instruction on how to progress a home exercise program. Participants will also need to complete a home exercise log.
  2. Education: Participants will be given homework to do at home in between online module sessions. Online quizzes will help review the educational material.
  Interventions: Other: Exercise; Other: Education
- Multi-visit, Physical Therapist Guided Rehabilitation (Active Comparator): Participants will attend 6 to 7 telehealth sessions over 8 weeks, which will last 30 to 45 minutes each and include:
  1. Exercise participation: Instruction from a physical therapist will be provided on how to complete a home exercise program between treatment sessions. Participants will also need to complete a home exercise log.
  2. Education: Participants will be given homework and online quizzes to do at home in between treatment sessions. The physical therapist will review the educational material at each visit.
  Interventions: Other: Exercise; Other: Education

INTERVENTIONS:
Other: Exercise — All participants will be instructed in a progressive Achilles tendon loading exercise program.
Other: Education — All participants will receive education on Achilles tendinopathy terminology, common symptoms, diagnosis, expected recovery timeline, importance of physical activity, self-management strategies, multiple factors influencing pain, alternative and adjunct treatment options.

SUMMARY:
This is a randomized controlled trial with individuals who have Achilles tendon pain. This study is designed to identify an effective rehabilitation program for Achilles tendon pain that expands access to care for military personnel and to predict treatment response. Limited or delayed access to healthcare can exacerbate the severity of pain and duration of disability due to AT. This is particularly relevant for individuals deployed to battlefield settings or are being seen in busy military treatment facilities. Therefore, it is crucial to identify efficient and effective treatment pathways that maximize healthcare access and facilitate a rapid and pain-free return to full duty.

DETAILED DESCRIPTION:
The objectives of this non-inferiority trial are to identify a rehabilitation program focused on education and exercise for AT that expands access to care for military personnel and to identify factors that predict responses to rehabilitation. The following aims will test our central hypothesis that a single-visit, PT-initiated rehabilitation program will be as effective in improving pain and reducing disability as a multi-visit, PT-guided rehabilitation program for AT and that within two weeks of initiating exercise treatment, early changes in patient-reported outcomes can identify responders.

Specific Aim 1. Determine the efficacy of a single-visit, PT-initiated rehabilitation program vs. a multi-visit, PT-guided rehabilitation program for AT.

Specific Aim 2. Identify early prognostic factors for individuals who experience the greatest improvement in pain and disability by four weeks.

Study Design. A single-blind, two-arm, parallel phase 2 randomized controlled trial is the study approach. Individuals with AT will be randomized to one of two rehabilitation programs: 1) self-guided intervention initiated with a single visit with a physical therapist (PT) via telehealth followed by modules that the participant can complete asynchronously, or 2) PT-guided intervention (standard of care) with six one-on-one telehealth visits. Study will enroll 160 individuals with AT across two sites (University of Iowa Hospitals & Clinics; Carl R. Darnall Army Medical Center, Fort Cavazos) and obtain baseline variables and immediate response at 2-weeks to characterize the sample. Outcomes will be assessed at 4 weeks (primary endpoint), 8 weeks, 26 weeks, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Pain localized to the Achilles tendon (insertion or midportion)
* AT pain greater than or equal to 3/10 with tendon-loading exercise

Exclusion Criteria:

* Younger than 18 years of age or older than 60 years of age
* BMI > 45 kg/m2
* Pain primarily due to a differential diagnosis, including paratendonitis, bursitis (retrocalcaneal or subcutaneous), posterior ankle impingement or os trigonum, irritation or neuropathy of the sural nerve, plantaris tendon involvement)
* Presence of a partial Achilles tendon tear or rupture on imaging or a history of Achilles tendon rupture that was verified by surgical or conservative management
* Attended physical therapy for AT in the past 3 months
* History of steroid injection to lower extremity tendons/fascia, ESWT or any injection to the Achilles tendon region in the past 3 months
* History of taking fluoroquinolones in the past 6 months
* History of surgery or invasive procedure for AT on side enrolling for treatment
* Diagnosed systemic conditions affecting the foot and ankle (e.g., rheumatoid arthritis, ankylosing spondylitis), endocrine disorder with complications (e.g., uncontrolled Type I or II diabetes, diabetic peripheral neuropathy), connective tissue disorder (e.g., Marfan's syndrome, Ehlers Danlos), or pregnancy
* At high risk for falls (four step square test >15 seconds)
* Refusal of randomization or unable or uninterested in completing virtual visits with a webcam or smart phone or completing quizzes and surveys

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Tendon Pain | From enrollment to 4 weeks
  Participants will report the intensity of movement-evoked pain during single limb heel raises using the Verbal Numeric Rating Scale (NRS, 0 to 10). Where "0" represents "no pain" and "10" indicates "worst pain imaginable."
Disability | From enrollment through 4 weeks
  Victorian Institute of Sports Assessment-Achilles (VISA-A) with score range from 0 to 100. A lower score indicates greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth L Chimenti, PT, PhD, Principal Investigator — University of Iowa; Matthew Frazier, PT, DPT, MS, ATC, Study Director — Carl R. Darnall Army Medical Center (CRDAMC), Fort Cavazos
Locations (2):
- United States (2):
  - University of Iowa Health Care - Gait Analysis Laboratory, Iowa City, Iowa
  - Carl R. Darnall Army Medical Center (CRDAMC), Fort Cavazos, Texas

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the Congressionally Directed Medical Research Programs Policy on Sharing Data and Research Resources, we will share the primary outcomes data and research resources, such as the rehabilitation handouts and videos. All data that is necessary to validate research outcomes and publications will be preserved and shared to allow other researchers the ability to reproduce the data and obtain additional findings that can advance the results. To ensure that other users can efficiently and accurately use the dataset, we will provide metadata and associated documentation. Information needed to understand the meaning of variable names and information about coding for missing data will be recorded in data dictionaries and readme files that will subsequently be shared alongside final datasets. Protocols, methods, statistical analyses, and any other relevant documentation
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available within 1 year of completing the study and remain available for at least 10 years
Access Criteria: A link to the data will be shared upon publication or within 1 year of completing the study, whichever occurs first. The primary outcome data and resources will be freely available to the public via Iowa Research Online repository. The repository is open access and maintained by the Libraries at the University of Iowa for the preservation and sharing of intellectual work of faculty, students, and staff.